CLINICAL TRIAL: NCT01759914
Title: Intraocular Pressure in Corticosteroid-treated Dermatology Patients
Brief Title: Ocular Pressure in Steroid-treated Dermatology Patients
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit sufficient number of subjects in required timeline.
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Yasaman Mansouri, MD, Specialist Registrar in Dermatology, University Hospitals Coventry and Warwickshire NHS Trust
Other Study IDs: YM076710
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Topical Corticosteroid-treated Dermatology Patients; Intra-ocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Potent topical steroid-treated: Patients treated with potent topical steroids
  Interventions: Drug: Potent topical steroid
- Superpotent topical steroid-treated: Patients treated with superpotent topical steroids
  Interventions: Drug: Superpotent topical steroid

INTERVENTIONS:
Drug: Potent topical steroid
  Groups: Potent topical steroid-treated
Drug: Superpotent topical steroid
  Groups: Superpotent topical steroid-treated

SUMMARY:
Ocular hypertension and glaucoma are eye conditions associated with abnormally high fluid pressure in the eye (called intraocular pressure or IOP). If left untreated, the elevated IOP may eventually cause damage to the nerve of the eye and potential impairment of vision.

The use of certain drugs has been identified as a risk factor for raised IOP, including various forms of administration of corticosteroids. Corticosteroids can also lead to cataract, which is clouding of the lens in the eye that can affect vision.

In this research study, we would like to find out whether the use of corticosteroids in our dermatology clinic leads to raised IOP, in order to identify patients at risk and to allow them to be more closely monitored than others. It is important to identify those patients who have a corticosteroid-induced pressure rise early enough to prevent them from permanent glaucomatous visual loss.

ELIGIBILITY:
Inclusion Criteria:

* patients on whom corticosteroid treatment is being introduced for a duration of at least 12 weeks

Exclusion Criteria:

* pregnant women
* patients already under glaucoma treatment
* patients unable to give informed written consent or those unable to cooperate fully with the assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dermatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure from baseline | after 1, 2 and 3 months
  Measurements will be done at 28 (+/- 7 days) days, 56 (+/- 7 days) days, and 90 (+/- 7 days)days after initiation of topical steroids.

SECONDARY OUTCOMES:
Whether there is any clinical evidence of cataract at the final visit of the study. | After 1, 2 and 3 months
  Measurements will be done at 28 (+/- 7 days) days, 56 (+/- 7 days) days, and 90 (+/- 7 days)days after initiation of topical steroids.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom